CLINICAL TRIAL: NCT04215770
Title: Comparison of Intravenous Co-amoxiclav Versus Benzyl Penicillin in Children With Severe Tonsillitis
Brief Title: Comparison of Intravenous Co-amoxiclav Versus Benzyl Penicillin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Combined Military Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Ahmed Khan, ENT consultant, Combined Military Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMH-01-2019
Record Dates: First submitted 2019-12-29; First posted 2020-01-02 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Tonsillitis Streptococcal
Keywords: Co-amoxiclav; Benzyl Penicilli; Tonsillitis
MeSH Terms: conditions — Tonsillitis

STUDY DESIGN:
Intervention Model Description: single blinded clinical trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inj Co-amoxiclav (Active Comparator): Group A children were advised Inj Co-amoxiclav 50 units/kg/day in 3 divided doses daily
  Interventions: Drug: inj co-amoxiclav 50 units/kg/day vs inj Benzyl Penicillin 25000 units/kg/day
- Inj Benzyl Penicillin (Active Comparator): Group B patients were advised inj Benzyl Penicillin 25000 units/kg/day in 3 divided doses
  Interventions: Drug: inj co-amoxiclav 50 units/kg/day vs inj Benzyl Penicillin 25000 units/kg/day

INTERVENTIONS:
Drug: inj co-amoxiclav 50 units/kg/day vs inj Benzyl Penicillin 25000 units/kg/day — Patients of both groups were examined and compared in terms of efficacy of treatment, safety and cost effectiveness
  Other Names: Group A and B

SUMMARY:
To compare intravenous Co-amoxiclav versus Benzyl penicillin in children with severe streptococcal tonsillitis in terms of efficacy, safety and cost effectiveness.

DETAILED DESCRIPTION:
Efficacy was measured through improvement (decrease in fever, settling lymphadenopathy and disappearance of tonsillar exudate) in Centor Criteria score on daily basis. Improvement i.e reduction in Centor Criteria score was recorded for all children till full recovery.

Safety was measured by frequency of hypersensitivity reactions or severe side effects of antibiotics necessitating stoppage of the drug. All the children in both Groups were given test dose of the antibiotic before giving full dose of antibiotic prescribed.

Cost effectiveness was compared in terms of total cost of injections (Co-amoxiclav versus Benzyl penicillin) which were administered to children in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Children who had 3 or 4 score according to Centor Criteria for tonsillitis/pharyngotonsillitis, were included in study
2. Children between ages of 5 to 15 years
3. Children with positive Rapid Antigen detection Test (RADT) for Streptococcus Pyogenes

Exclusion Criteria:

1. Immunocompromised children
2. Children with known hypersensitivity to Penicillins (esp Coamoxiclav and Benzyl penicillin)
3. Children with liver or renal failure
4. Children who were already using any oral or parenteral antibiotics

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 310 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
treatment efficacy | 10 days
  full recovery (Centor score became zero/nil)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Khan, MBBS, FCPS, Principal Investigator — CMH Mardan
Locations (1):
- CMH Mradan, Mardan, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No
It will not be shared